CLINICAL TRIAL: NCT06084949
Title: Effect of Nordic Walking and Inspiratory Muscle Training to Promote Cardiopulmonary Function in Patients With Knee Osteoarthritis
Brief Title: Effect of Structured Exercise in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20230703001
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee; Physical Inactivity
Keywords: exercise; pain; function
MeSH Terms: conditions — Osteoarthritis, Knee; Sedentary Behavior; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated into intervention group or controlled group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor won't know the allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic walking group or inspiratory muscle training (Experimental): In experimental group, investigator will coordinate with the patients with mild-to-moderate knee osteoarthritis to take the Nordic walking, while the patients with end-stage knee osteoarthritis to take inspiratory muscle training. All participants are required to maintain their daily activities and routine management.
  Interventions: Device: Nordic walking or inspiratory muscle training
- Control group (No Intervention): In control group, participants are required to maintain their daily activities and routine management.

INTERVENTIONS:
Device: Nordic walking or inspiratory muscle training — Nordic walking is a form of low-impact aerobic exercise that incorporates the use of walking poles. And inspiratory muscle training is a type of exercise that provides resistance during the inhalation phase.
  Arms: Nordic walking group or inspiratory muscle training

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effect of Nordic walking and inspiratory muscle training (IMT) on cardiopulmonary function in patients with knee osteoarthritis (OA). Mild-to-moderate knee OA patients are randomly allocated into Experimental group (Nordic walking plus routine management) or Control group (Routine management). While End-stage knee OA patients are randomly allocated into Experimental group (IMT plus pre-operative rehabilitation exercise) or Control group (Pre-operative rehabilitation exercise). Participants are invited to undergo two assessments, including baseline assessment, post-intervention assessment. Researchers will compare two groups to see if the cardiopulmonary function can be improved after intervention.

DETAILED DESCRIPTION:
This study recruits patients with different stages and assigns them into different interventions and comparing the effect with those not receiving intervention. It will provide the evidence in terms of the exercise that can promote cardiopulmonary function and at the same time reduce pain and disability for patients with different stages of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* pain on the most days in one or both knees in the past month;
* difficulty with at least one of daily living activities measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale;
* radiographic evidence of knee OA in the tibial-femoral compartment (Kellgren and Lawrence grade, K/L ≥1, K/L 1-3 regarded as mild-to-moderate knee OA, others waiting for knee arthroplasty regarded as end-stage knee OA);
* with normal or corrected visual and auditory function and walking unaided;
* primary knee OA for more than 6 months, be stable on medication for at least 3 weeks.

Exclusion Criteria:

* knee surgery priorly;
* have steroid injection in previous three weeks;
* have inflammatory arthritis (e.g., rheumatoid); or unstable angina, or myocardial infarction, or cardiac surgery; or stroke; or treatment with steroids, hormones, or cancer chemotherapy; or pulmonary diseases (force vital capacity<80% of predicted and/or forced expiratory volume at first second<70% of predicted); or a history of exercise-induced asthma;
* unable to understand the procedure and potential risks of the study;
* medically unstable that indicate unsafe to participate in exercise test

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The six-minute walk test | Baseline, up to 8 weeks
  Cardiopulmonary function
30-sec chair stand test | Baseline, up to 8 weeks
  Cardiopulmonary function
Grip strength | Baseline, up to 8 weeks
  Cardiopulmonary function
Timed up-and-go test | Baseline, up to 8 weeks
  Cardiopulmonary function
Quadriceps strength | Baseline, up to 8 weeks
  Cardiopulmonary function

SECONDARY OUTCOMES:
Forced vital capacity | Baseline, up to 8 weeks
  Pulmonary function
Forced expiratory volume at first second | Baseline, up to 8 weeks
  Pulmonary function
Maximum voluntary ventilation | Baseline, up to 8 weeks
  Pulmonary function
Inspiratory muscle strength | Baseline, up to 8 weeks
  Pulmonary function
Inspiratory muscle endurance | Baseline, up to 8 weeks
  Pulmonary function
Quadriceps muscle oxygenation | Baseline, up to 8 weeks
  Quadriceps muscle function
Multidimensional Fatigue Inventory | Baseline, up to 8 weeks
  Total scores range from 20-100, , the higher scores indicating a higher level of fatigue.
Medical Research Council scale | Baseline, up to 8 weeks
  Total scores range from 0-4, the higher scores indicating a higher level of dyspnea.
Physical Activity Scales for the Elderly | Baseline, up to 8 weeks
  Total scores range from 0-793, the higher scores indicating a higher level of physical activity.
Actigraph | Baseline, up to 8 weeks
  Physical activity level
Pittsburgh Sleep Quality Index | Baseline, up to 8 weeks
  Total scores range from 0-21, '0' indicating no difficulty and '21' indicating severe difficulties in all areas.
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline, up to 8 weeks
  Knee-related symptoms and function, total scores range from 0-96, the higher scores indicating the worse symptom and function.
12-Item Short Form Health Survey | Baseline, up to 8 weeks
  Total scores range from 0-100, the higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Amy FU, PhD, Principal Investigator — Department of Rehabilitation Sciences
Locations (1):
- The Hong Kong Polytechnic University, Kowloon City, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.